CLINICAL TRIAL: NCT06433154
Title: Arthroscopic Lysis and Lavage in Patients With Internal Derangement of the Temporomandibular Joint: A Retrospective Cohort Study on Jaw Mobility, Pain and Health-related Quality of Life
Brief Title: Arthroscopy of the Temporomandibular Joint. On Jaw Mobility, Pain and HRQoL
Status: Completed | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 230_20211018_073
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Arthroscopic Surgery; Temporomandibular Joint; Health-Related Quality Of Life; Follow-Up Studies; Observational
Keywords: Arthroscopy; TMJ; PROM; HRQoL
MeSH Terms: interventions — Arthroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthroscopic surgery to the temporomandibular joint: Arthroscopic lysis and lavage in patients with internal derangement of the temporomandibular joint. Retrospective observational follow-up cohort trial.
  Interventions: Procedure: Arthroscopic surgery

INTERVENTIONS:
Procedure: Arthroscopic surgery — Arthroscopic treatment (lysis and lavage) of internal derangement of the temporomandibular joint.

SUMMARY:
The aim of the present study is to retrospectively investigate whether arthroscopic treatment in patients with TMD symptoms depending on internal derangement of the temporomandibular joint (TMJ) gives a satisfying result on the patient's quality of life.

Based on previous studies it is hypothesized that patients suffering from TMD depending on internal derangement would through Patient Reported Outcome Measures (PROM) evaluate the treatment efficacy from an arthroscopic treatment as a benefit to their quality of life.

Further, the study intends to find out if the patient reported outcome measures (PROM) on health-related quality of life (HRQoL) outcome correlates with clinical follow-up measures after arthroscopic treatment of internal derangement of the temporomandibular joint.

The primary objective is to measure the correlation between the results from a HRQoL questionnaire and mouth opening. Secondary, the effect of mouth opening on HRQoL is being explored.

The primary prediction variable is the surgical treatment. Outcome variables are treatment evaluation quality of life (PROM) based on a validated questionnaire; Jaw Functional Limitation Scale (JFLS), age, gender, time from diagnosis to treatment, severity of symptoms (pain, mouth opening ability) and time from treatment to evaluation.

DETAILED DESCRIPTION:
Sample Patients that on referral and examination in 2006 to 2019 at the department of Oral and Maxillofacial Surgery, Skåne University Hospital (SUS) was diagnosed with Temporo Mandibular dysfunction (TMD), will be recruited for participation in the study. Patients aged over 20 years with a dysfunction presenting painful clicking or locking of the Temporomandibular Joint (TMJ), that underwent an arthroscopic treatment the TMJ on one side will be asked for a follow-up. The indication for surgical treatment of these patients was anterior disc displacement combined with pain or "Closed Lock" (disc displacement without reduction). The clinical classification is based on general medical history, history of dysfunction (debut, duration, frequency, character, diurnal variation, symptoms relief, symptoms accentuation), clinical recordings (muscle palpation, joint palpation, recordings of jaw movements and provocation maneuvers, eg Krogh-Poulsen test). The referred patients with TMD were, before selected to arthroscopic treatment, separated into joint associated TMD or muscular associated TMD. Patients with only muscular or mainly muscular symptoms were excluded from arthroscopic treatment and were offered alternative treatment. An important measurement for this selection is the Krogh-Poulsen test. The surgical treatment was carried out by three Oral and Maxillofacial surgeons with equal clinical experience. The sample was during the study period equally distributed between the surgeons. Patients with generalized joint disease, previous surgical treatment in the TMJ, less than 12 months of follow up time and/or had additional surgical treatment during the study period will be excluded from the study.

Surgical Method Surgical approach to the TMJ was established through a transcutaneous preauricular stab entry with a sharp 1,9 mm trocar (KARL STORZ SE & Co. KG, Tuttlingen, Germany) to the upper joint compartment. A second entry was made with a 1 mm syringe for drainage of the saline solution used for lavage of the upper joint compartment through the trocar cannula. Arthroscopic inspection and visual recording of the upper joint compartment was performed with an optical instrument placed through the trocar cannula. The optical instrument was replaced by a blunt tip, which was used for releasement of adherences between the joint surfaces, as well as stretching of the synovia (lysis). The upper joint compartment was flushed with a minimum of 200ml saline solution (lavage). Finally 1 ml morphine 10 mg/ml was injected through the drainage syringe for postoperative pain relief. Postoperatively the patient was instructed in a jaw mobility training programme, NSAID's (Ibuprofen 400mg orally every 6 to 8 hours) and jaw rest (not to chew) for at seven to thirty days. The duration of the postoperative regime was decided at weekly follow-ups.

Variables The primary prediction variable is the surgical treatment. The primary outcome variable is a treatment evaluation quality of life questionnaire score, based on a validated questionnaire; Jaw Functional Limitation Scale (JFLS). The questionnaire will be tested for reliability through repeated recording with at least 2 months gap between for 30 of the patients. Other predictor variables that could affect the treatment outcome are age, gender, time from diagnosis to treatment, severity of symptoms (pain, mouth opening ability), time from treatment to evaluation, postoperative jaw mobility and improvement of jaw mobility. After the patients have been consented for the study, they will be asked to fill in the Patient Reported Outcome Measures (PROM) questionnaire on self-perceived jaw function (JFLS). The questionnaire will be sent out to all included patients during 2022.

Retrospectively, the following data will be recorded from patient records: gender, age (at surgery), jaw movements, pain, pre surgical diagnosis (clinical) and surgical diagnosis (arthroscopic).

Statistical methods The sample size is based on a total number of 500 patients to be recruited for the enquiry study. In addition, 4000 patients will be included for analysis of journal records alone. Analysis will use mean values, confidence intervals, standard deviations, the Cox regression for evaluation of clinical records treatment outcome and logistic regression for the PROM evaluation. Differences in mouth opening and pain scores, preoperatively and postoperatively will be compared with McNemar's test.

Wilcoxon's paired-sample test will be used for analyzing mouth opening before and after surgery as a numeric variable. Mann-Whitney-test will be used to detect differences between questionnaire responses and clinical findings, i.e. pain and mouth opening. The limit for significant difference will be set to p=0.05. Two-sided p-values will be used. A correlation analysis (Spearman) for postoperative mouth opening and JFLS-score, and progression of mouth opening and JLFS-score will be used.

ELIGIBILITY:
Inclusion Criteria:

Patients referred to the Department of Oral and Maxillofacial Surgery, Lund University Hospital between 2006 to 2019 with a temporomandibular dysfunction presenting painful clicking or locking of the TMJ and has underwent an arthroscopic treatment the TMJ on one side.

Patients aged over 20.

Exclusion Criteria:

Patients with only muscular or mainly muscular originated TMJ symptoms. Present generalized joint disease, previous surgical treatment in the TMJ, less than 12 months of follow up time and patients which have had additional surgical treatment during the study period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients which had surgical treatment, were anterior disc displacement combined with pain or "Closed Lock" (disc displacement without reduction).
  Patients aged over 20.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Jaw mobility | At least one year follow-up after surgery.
  Measured range of mandibular movements.

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQoL) | At least one year follow-up after surgery.
  Patient reported outcome measure with a HRQoL questionaire.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bengtsson, DDS, PhD, Principal Investigator — Lund University Hospital
Locations (2):
- Sweden (2):
  - Dept Oral and Maxillofacial Surgery, Lund
  - Martin Bengtsson, Lund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bengtsson M, Fransson P. Do patient-reported outcome measures correlate with clinical follow-up after arthroscopic treatment of internal derangement of the temporomandibular joint? J Stomatol Oral Maxillofac Surg. 2021 Sep;122(4):e21-e26. doi: 10.1016/j.jormas.2021.03.003. Epub 2021 Apr 9. PMID 33845189